CLINICAL TRIAL: NCT04747938
Title: Treating Frozen Shoulder With Integrative Medicine Approach by the Energy Accumulator - a Prospective Clinical Trial
Brief Title: Frozen Shoulder Treated by Energy Accumulator
Acronym: FShouEnAcc
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Ho Ki Wai, Clinical Professional Consultant, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014.092-T
Record Dates: First submitted 2021-02-05; First posted 2021-02-10 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-07

CONDITIONS: Frozen Shoulder
Keywords: Frozen Shoulder; Integrative Medicine; Energy Accumulator
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Energy accumulator (Experimental): Energy Accumulator was a portable handheld device invented for local heat therapy for healthcare purpose. All subjects treated with thermal therapy using the Energy Accumulator by acupoint concepts.
  Interventions: Device: Energy accumulator
- Home exercise program (Experimental): Home exercises aimed at providing gentle mobilization at the shoulder and were capable of carrying out at home. Patients were requested to perform the movements on a daily basis within the first 4 weeks of treatment. Four movements were involved: Movement 1 - Pendular Exercise, Movement 2 - Circle Exercise, Movement 3 - Wall Climbing Exercise, and Movement 4 - Lie on bed and move both arms up and down.
  Interventions: Behavioral: Home exercise program

INTERVENTIONS:
Device: Energy accumulator — All subjects treated with thermal therapy using the Energy Accumulator by acupoint concepts. The course included 8 sessions of treatment, twice every week for 4 weeks. Each session lasted for 30-45 minutes. During heat therapy, the ceramic nozzle of the Energy Accumulator was lightly pressed in contact of the skin, without any contact medium, and moved slowly along the meridians with some circular movements.
  Arms: Energy accumulator
Behavioral: Home exercise program — Home exercises aimed at providing gentle mobilization at the shoulder and were capable of carrying out at home. Patients were requested to perform the movements on a daily basis within the first 4 weeks of treatment. Four movements were involved: Movement 1 - Pendular Exercise, Movement 2 - Circle Exercise, Movement 3 - Wall Climbing Exercise, and Movement 4 - Lie on bed and move both arms up and down.
  Arms: Home exercise program

SUMMARY:
Frozen shoulder is a painful and disabling disorder of unclear cause, affecting middle-age people after their 5th decades. They suffer from annoying pain and limited shoulder mobility. Energy Accumulator provides a better way of relief through an integrative medicine concept.

DETAILED DESCRIPTION:
Frozen shoulder is common among middle-aged persons in the 5th and 6th decades. The pain can be acute or chronic. Patients feel stiffness over the shoulder, shown by restriction in range of motion. The etiology includes trauma, cervical disc degeneration, physical strain, psychosocial problems and even genetic factors. The predisposing factors include immobilization of the arm for a long time, rotator cuff or biceps tendinitis, tenosynovitis of the long head of the biceps, congenital deformity of the shoulder girdle, scapula-costal cementing, ligamentous injury, osteoarthritis, muscular fibrosis or nutritional deficiencies. The pathology is unclear but it is widely believed that it is related to inflammation in the joint and surrounding soft tissues which lead to fibrosis. Frozen Shoulder can be divided into Primary Frozen Shoulder which occurs spontaneously without other diseases; and Secondary Frozen Shoulder is associated with joint diseases, such as osteoarthritis or fractures.

UKFROST was a multi-centre randomized clinical trial comparing 3 parallel groups (arms) of frozen shoulder patients treated 1) under anaesthesia + steroid injection 2) under anaesthesia + arthoscopy, and 3) physiotherapy + steriod injection..The large-scale study proves physiotherapy program beneficial to frozen shoulder patients, and, the effectiveness might further improve by introducing East-Meets-West component - Chinese Medicine.

ELIGIBILITY:
Inclusion Criteria:

* male or female gender with age between 40-65
* affect one shoulder only
* onset is more than 3 months at the time of inclusion into the study

Exclusion Criteria:

* unstable medical conditions
* unstable mental state
* have skin lesion over the shoulder
* skin sensitivity to heat
* pregnant or under lactation
* could not comply with heat treatment of the shoulder.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2015-08-03 (Actual); Study Completion 2015-10-24 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (10-point Likert scale) | Baseline
  A pain scale containing integers between min 0 and max 10. The higher scale the better outcome (less pain)
Visual Analogue Scale (10-point Likert scale) | 4 weeks
  A pain scale containing integers between min 0 and max 10. The higher scale the better outcome (less pain)
Oxford Shoulder Score (OSS) | Baseline
  12-item patient-reported patient reported outcome specifically designed and developed for assessing outcomes of shoulder surgery e.g. for assessing the impact on patients' quality of life of degenerative conditions such as arthritis and rotator cuff problems. Min 0 Max 48. The higher score the better outcome.
Oxford Shoulder Score (OSS) | 4 weeks
  12-item patient-reported patient reported outcome specifically designed and developed for assessing outcomes of shoulder surgery e.g. for assessing the impact on patients' quality of life of degenerative conditions such as arthritis and rotator cuff problems. Min 0 Max 48. The higher score the better outcome.
Shoulder Pain and Disability Index (SPADI) | Baseline
  (SPADI) is a self-administered questionnaire that consists of two dimensions, one for pain and the other for functional activities. Min 0 Max 100. The lower the better outcome.
Shoulder Pain and Disability Index (SPADI) | 4 weeks
  (SPADI) is a self-administered questionnaire that consists of two dimensions, one for pain and the other for functional activities. Min 0 Max 100. The lower the better outcome.
Short Form-12 (SF-12) | Baseline
  SF-12 is a self-reported outcome measure assessing the impact of health on an individual's everyday life. Min 0 Max 100. The higher scores the better outcome.
Short Form-12 (SF-12) | 4 weeks
  SF-12 is a self-reported outcome measure assessing the impact of health on an individual's everyday life. Min 0 Max 100. The higher scores the better outcome.

OTHER OUTCOMES:
Range of motion | Baseline
  To measure the range of motion of the affected and unaffected shoulder. Min 0 Max 180 degrees. The higher number the better.
Range of motion | 4 weeks
  To measure the range of motion of the affected and unaffected shoulder. Min 0 Max 180 degrees. The higher number the better.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Ki-Wai Ho, Dr., Principal Investigator — Chinese Univerisity of Hong Kong

IPD SHARING:
Plan to Share IPD: No